CLINICAL TRIAL: NCT06705647
Title: Analyzing Acoustic Properties of the Vowel "a" Collected Via Mobile Phone From Individuals Diagnosed With Chronic Obstructive Pulmonary Disease and Health Control Groups
Status: Active, not recruiting | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Excellence Center at Linköping - Lund in Information Technology (ELLIIT) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BTH-6.1.1-0198-2024
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acoustic features; Statistic analysis; Mel frequency cepstral coefficients; Vowel quadrilateral
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: 24 COPD participants, 12 Female and 12 Male.
  Interventions: Other: Chronic Obstructive Pulmonary Disease (COPD)
- HC: 24 HC participants, 12 Female and 12 Male.
  Interventions: Other: Chronic Obstructive Pulmonary Disease (COPD)

INTERVENTIONS:
Other: Chronic Obstructive Pulmonary Disease (COPD) — The base line acoustic and mel frequency ceprtum coefficients will be analysed statistically between COPD voices and healthy control groups to highlight the correlation between COPD and its effects on voice production.
  Other Names: Healthy Control (HC)

SUMMARY:
The Study aims to identify the changes in voice caused by Chronic Obstructive Pulmonary Disease (COPD) statistically for identifying the potential digital voice biomarkers.

DETAILED DESCRIPTION:
1058 voice recordings collected via mobile phones over time in form of the Swedish utterance of vowel "a" will be analysed using vowel quadrilateral space and the Mann-Whitney U test.

The significance threshold p-value will be set to 0.05, and vocal features consisting of 101 base line acoustic features and MFCC features will be analysed between the COPD and HC groups. The most significant features that remain under the significance threshold will be reported.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old and older.

Exclusion Criteria:

* being under 18 years old and older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data collected from participants 18 years old and older with and without COPD diagnosis will be used. The participants will be balanced on a gender and age basis.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Acoustic Voice Features Between COPD and Healthy Control Participants Difference in Acoustic Voice Features Between COPD and Healthy Control Participants | 30 weeks
  This study assesses differences in baseline acoustic features (e.g., F0, HNR, jitter, shimmer, and formant frequencies), MFCC features (1-13 and derivatives Δ, ΔΔ), and vowel quadrilateral metrics (VSA from F1 and F2 of the sustained vowel 'a') between COPD and healthy controls. Acoustic features are extracted using Parselmouth and Praat, while MFCC features are computed with Librosa. Descriptive statistics (median, mean, std) are calculated, and group differences are tested for significance using the Mann-Whitney U test. Units include median, mean, std for each feature and VSA (Hertz²). Results will include p-values for group comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: No
Participant data can not be shared due to the GDPR. However, the dataset created can be available upon request from the institution.

REFERENCES:
- [Derived] Idrisoglu A, Moraes ALD, Cheddad A, Anderberg P, Whitling S, Jakobsson A, Berglund JS. Feature Analysis of the Vowel [a:] in Individuals With Chronic Obstructive Pulmonary Disease and Healthy Controls. J Voice. 2025 Oct 29:S0892-1997(25)00429-1. doi: 10.1016/j.jvoice.2025.10.013. Online ahead of print. PMID 41168019